CLINICAL TRIAL: NCT06425276
Title: A Multicenter, Open-Label, Safety and Efficacy Study of High Dose Melphalan Hydrochloride for Injection for Myeloablative Conditioning in Multiple Myeloma Patients Undergoing Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Evaluate Safety and Efficacy of High-dose Melphalan HCL for Injection in MM Patients With Auto-HSC Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CASI Pharmaceuticals (China) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVOM-CL-001
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- High-dose Melphalan HCl for Injection treatment arm (Experimental): Patients will receive Melphalan HCl for Injection dosed at 100 mg/m2 on Day -3 and Day -2. Following 1 day of rest after the myeloablative conditioning (Day -1), patients will receive an autologous graft with a minimum cell dose of 2 × 106 CD34+ cells/kg of patient body weight (Day 0).
  Interventions: Drug: Melphalan Hydrochloride for Injection

INTERVENTIONS:
Drug: Melphalan Hydrochloride for Injection — During the Study Period, patients will receive Melphalan HCl for Injection dosed at 100 mg/m2 on Day -3 and Day -2.
  Other Names: Evomela

SUMMARY:
The goal of this clinical trial is to learn if high-dose Melphalan HCl for Injection works to treat multiple myeloma. It will also learn about the safety of high dose Melphalan HCl for Injection. The main questions it aims to answer are:

Does high-dose Melphalan HCl for Injection deplete bone marrow activity which results in a better outcome of patients'own stem cell (blood-forming cell) transplantation? What medical problems do participants have when taking high-dose Melphalan HCl for Injection? How fast is the high-dose Melphalan HCl for Injection cleared out from blood?

Participants will:

* Take high-dose Melphalan HCl for Injection for 2 days
* Have stem cell transplantation one day after treatment
* Stay in the hospital for at least 10days and visit the clinic once every week for the first month after transplantation and every month after for checkups and tests.

DETAILED DESCRIPTION:
Autologous stem cell transplantation (ASCT) is a standard of care in transplant-eligible MM patients which has been demonstrated with a better complete remission rate (CR) and with longer survival. High-dose melphalan (200 mg/m2) has been the most commonly used conditioning regimen for ASCT in MM. EVOMELA (melphalan HCl for Injection) stabilized with Captisol, a specially modified cyclodextrin, has been believed to have better solubility and stability upon reconstitution which result in decreased toxicity, increased convenience and flexibility of administration without comprising efficacious data. Melphalan HCl for Injection has been approved by NMPA as a standard conditioning drug for ASCT in MM patients. The current study evaluated the efficacy, safety, and PK profile for high-dose Melphalan HCl for Injection as a myeloablative conditioning regimen in Chinese symptomatic transplant-eligible MM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as symptomatic multiple myeloma, according to the International Myeloma Working Group's IMWG Guidelines for the Diagnosis and Treatment of Multiple Myeloma, treatment is necessary and suitable for autologous hematopoietic stem cell transplantation;
2. When signing the informed consent form, males and females aged ≥ 18 years and ≤ 65 years old;
3. Adequate autologous hematopoietic stem cells were collected, defined as peripheral blood stem cells containing at least 2 x 106 CD34+cells/kg that have not been manipulated or refrigerated;
4. Important organ functions meet the following conditions:

   i. Echocardiography indicates left ventricular ejection fraction (LVEF) ≥ 40%;

   ii. Serum total bilirubin<2 times the upper limit of normal value, alanine aminotransferase (ALT) and aspartate aminotransferase (AST)<3 times the upper limit of normal value;

   Iii. creatinine clearance rate>60 mL/min ;

   Iv. Blood oxygen saturation>92% in non oxygenated state, without significant ventilation or ventilation dysfunction;
5. The Eastern Oncology Collaborative Group (ECOG) physical fitness status of the subjects is 0, 1, or 2;
6. The subject or their legal guardian voluntarily signs an informed consent form approved by the ethics committee before participating in the study, and agrees to complete the entire study treatment according to the clinical trial protocol.

Exclusion Criteria:

1. Multiple myeloma subjects without treatment indications;
2. Suffering from plasma cell leukemia;
3. Suffering from systemic amyloidosis;
4. Subjects with extramedullary plasma cell tumors did not reach PR after induction therapy;
5. Suffering from POEMS syndrome (multiple peripheral neuropathy, organ enlargement, endocrine disorders, M-proteinemia, skin changes);
6. Suffering from Fahrenheit macroglobulinemia;
7. Subjects with non secretory multiple myeloma;
8. Subjects with active bacterial, viral, or fungal infections who require oral or intravenous antibiotic treatment according to the researcher's judgment;
9. The expected survival period of the subjects is less than 6 months;
10. Previously suffering from other malignant tumors, except for cured basal cell carcinoma or cervical carcinoma in situ. Malignant tumors that have undergone curative treatment and achieved complete remission (CR) for more than 5 years can be enrolled. If malignant tumors receive curative treatment but have achieved complete remission (CR) for ≤ 5 years, they cannot be enrolled unless approved by the sponsor;
11. Pregnant or lactating women;
12. Subjects who have fertility and are unwilling to take appropriate contraceptive measures within 3 months after signing the informed consent form until the end of treatment in this study;
13. Positive for human immunodeficiency virus (HIV) antibodies;
14. Subjects with positive hepatitis B virus DNA;
15. The subject receives other concurrent anti-tumor treatments (including chemotherapy, radiation therapy, hormone therapy, or immunotherapy) within 30 days prior to autologous hematopoietic stem cell transplantation, or plans to receive any such treatments before the last study visit on day 95 ± 5;
16. The side effects of chemotherapy drugs received before administration have not yet recovered, defined as not regressing to level 0/1 of the National Cancer Institute's Common Terminology Standard for Adverse Events (NCI-CTCAE v5.0), or at the level specified in the inclusion/exclusion criteria, except for adverse events such as hair loss that the researcher assessed and deemed not to affect the safety of the subject's participation in this study;
17. Allergy or intolerance to any component of the investigational drug formulation;
18. Participants participate in other clinical trials within one month before signing the informed consent form;
19. According to the researcher's judgment, subjects who are not suitable for enrollment, may affect treatment evaluation, or are at inappropriate risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-09-18 (Actual)

PRIMARY OUTCOMES:
Rate of patients achieveing myeloablation | 95±5 days after ASCT
  To record the percentage of patients who achieve myeloablation which is defined as absolute neutrophil count [ANC] <0.5 × 109/L, absolute lymphocyte count [ALC] <0.1 × 109/L, or platelet count <20,000/mm3 in 2 consecutive daily assessments.
Time to achieveing myeloablation | 95±5 days after ASCT
  To record the time, in days, from the date of first dose of High-dose Melphalan HCL for Injection to the date of myoloablation which is defined as absolute neutrophil count [ANC] <0.5 × 109/L, absolute lymphocyte count [ALC] <0.1 × 109/L, or platelet count <20,000/mm3 in 2 consecutive daily assessments.
Time to achieveing neutrophil engraftment | 95±5 days after ASCT
  To record the time, in days, from the date of Auto-HSCT to the date when absolute neutrophil count (ANC) >0.5 × 109/L in 3 consecutive daily assessments.
Time to achieving platelet engraftment | 95±5 days after ASCT
  To record the time, in days, from the date of Auto-HSCT to the date when untransfused platelet measurement >20,000/mm3 in 3 consecutive daily assessments.
Incidence of Treatment-related Motality (TRM) | 95±5 days after ASCT
  To characterize the safety, tolerability of High-dose Melphalan HCL for Myeloablation in MM Patients With Auto-HSC Transplantation by recording the incidence of death without relapse or progression of the disease.
Incidence and severity of AEs and SAEs, including changes in laboratory values | 95±5 days after ASCT
  To characterize the safety, tolerability of High-dose Melphalan HCL for Injection for Myeloablation in MM Patients With Auto-HSC Transplantation.

SECONDARY OUTCOMES:
Overall Response (ORR) | 95±5 days after ASCT
  Response assessment per International Myeloma Working Group (IMWG) criteria
Tmax of Melphalan HCL for Injection derived from plasma concentrations | 24 Hours
  Tmax of Melphalan HCL for Injection derived from plasma concentrations of each administration
T1/2 of Melphalan HCL for Injection derived from plasma concentrations | 24 Hours
  T1/2 of Melphalan HCL for Injection derived from plasma concentrations of each administration
Cmax of Melphalan HCL for Injection derived from plasma concentrations | 24 Hours
  Cmax of Melphalan HCL for Injection derived from plasma concentrations of each administration
AUC of Melphalan HCL for Injection derived from plasma concentrations | 24 Hours
  AUC of Melphalan HCL for Injection derived from plasma concentrations of each administration

CONTACTS AND LOCATIONS:
Overall Officials: Kaiyan Liu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No